CLINICAL TRIAL: NCT01450774
Title: A Single Centre, Randomised, Double-blind, Double-dummy, 2-way Cross Over Study to Compare Safety Assessed by Knemometry and Urinary Cortisol Measurements of CHF1535 50/6 Pmdi (Fixed Combination of Beclomethasone Dipropionate and Formoterol Fumarate) and the Free Combination of Licensed Beclomethasone Dipropionate and Formoterol Fumarate in Asthmatic Children Already Treated With Inhaled Corticosteroids
Brief Title: Comparison of Combination of Beclomethasone Dipropionate and Formoterol Fumarate Versus Single Components Assessed by Knemometry and Urinary Cortisol Measurements in Asthmatic Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1012-PR-0051
Record Dates: First submitted 2011-09-23; First posted 2011-10-12 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Childhood Asthma
MeSH Terms: interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 1535 50/6µg (Experimental)
  Interventions: Drug: CHF 1535 50/6µg
- beclomethasone dipropionate 50µg + formoterol fumarate 6µg (Active Comparator)
  Interventions: Drug: beclomethasone dipropionate 50µg + formoterol fumarate 6µg

INTERVENTIONS:
Drug: CHF 1535 50/6µg — fixed combination of beclomethasone dipropionate 50µg + formoterol fumarate 6µg
  Arms: CHF 1535 50/6µg
Drug: beclomethasone dipropionate 50µg + formoterol fumarate 6µg — free combination of beclomethasone dipropionate 50µg + formoterol fumarate 6µg
  Arms: beclomethasone dipropionate 50µg + formoterol fumarate 6µg

SUMMARY:
This is a single centre, double-blind, double-dummy, randomised, single-centre, 2-way cross-over study in asthmatic children already treated with inhaled corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Prepuberal male and female outpatients, ≥ 5 and ≤ 11 years old in Tanner stadium I according to Investigator's assessment
* Clinical diagnosis of mild asthma during at least two months prior to screening visit
* Forced Expiratory Volume during the first second (FEV1) > 80% of predicted normal values at screening visit

Exclusion Criteria:

* Endocrinological diseases including growth impairment or other chronic diseases
* Any concomitant disease requiring additional treatment with topic or systemic glucocorticosteroids

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Lower leg growth rate measured by knemometry | after a 2 week treatment

SECONDARY OUTCOMES:
24-hour urinary free cortisol/creatinine levels | after a 2 week treatment period
Changes in pre-dose morning and evening PEF (L/min) | pre and after a 2 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hans Bisgaard, MD, Principal Investigator — BørneAstmaKlinikken
Locations (1):
- BørneAstmaKlinikken, Copenhagen, Denmark

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-023637-29